CLINICAL TRIAL: NCT01813630
Title: Phase III Clinical Trial for Assessment of Efficacy and Safety of DA-3002 (Recombinant Human Growth Hormone) in Patients With Turner's Syndrome
Brief Title: A Clinical Study to Assess the Efficacy and Safety of DA-3002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA3002_TS_III
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Turner's Syndrome
Keywords: Turner's Syndrome; Short Stature; Dwarfism
MeSH Terms: conditions — Turner Syndrome; Dwarfism | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA-3002 (Experimental): 0.14 IU (0.045-0.050mg)/kg/day of DA-3002 is injected for 52 weeks by changing injecting areas
  Interventions: Drug: DA-3002
- Genotropin® (Active Comparator): 0.14 IU (0.045-0.050mg)/kg/day of Genotropin is injected for 52 weeks by changing injecting areas
  Interventions: Drug: Genotropin®

INTERVENTIONS:
Drug: DA-3002
  Arms: DA-3002
Drug: Genotropin®
  Arms: Genotropin®

SUMMARY:
A study demonstrates the non-inferiority of DA-3002 when compared with Genotropin®.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Turner's Syndrome through chromosome analysis
* The chronological age: 2≤AGE≤12
* The yearly growth rate should be less than 6cm; the bone age should be equal or less than 12; the height ≤ 10th percentile for the heights of their agemates
* Before the adolescence, Tuner stage I (breast)
* Normal thyroid function

Exclusion Criteria:

* Growth hormone was administered for 12 months or longer in the past
* Treated with estrogen or adrenal androgens for 12 months or longer in the past
* Malignancy, CNS Trauma, Psychiatric Disorder

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Annualized height velocity(cm/year) after 52 weeks | 52 weeks
  Height velocity calculated with height measured at Baseline and after 52 weeks was converted to annual growth rate

SECONDARY OUTCOMES:
Changes in height standard deviation score after 52 weeks | 52 weeks
Changes in bone maturation(changes in bone ages/changes in chronological age) | 52 weeks
Changes in IGF-1 | 52 weeks
Changes in IGFBP-3 | 52 weeks

OTHER OUTCOMES:
Changes in anti-growth hormone antibody | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Han Wook Yoo, M.D., Ph.D., Principal Investigator — Asan Medical Center; Byung Kyu Suh, M.D., Ph.D., Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea; Cheol Woo Ko, M.D., Ph.D., Principal Investigator — Kyungpook National University Hospital; Kee Hyoung Lee, M.D., Ph.D., Principal Investigator — Korea University Anam Hospital; Dong Kyu Jin, M.D.,Ph.D., Principal Investigator — Seoul Medical Center; Choong Ho Shin, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Jin Soon Hwang, M.D., Ph.D., Principal Investigator — Aju University Hospital; Ho Seong Kim, M.D., Ph.D., Principal Investigator — Severance Children's Hospital Yonsei University; Woo Young Jeong, M.D., Ph.D., Principal Investigator — Pusan University Hospital; Chang Jong Kim, M.D., Ph.D., Principal Investigator — Chonnam National University Hospital; Heon Suk Han, M.D., Ph.D., Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim J, Kim MS, Suh BK, Ko CW, Lee KH, Yoo HW, Shin CH, Hwang JS, Kim HS, Chung WY, Kim CJ, Han HS, Jin DK. Recombinant growth hormone therapy in children with Turner Syndrome in Korea: a phase III Randomized Trial. BMC Endocr Disord. 2021 Dec 10;21(1):243. doi: 10.1186/s12902-021-00904-5. PMID 34893062